CLINICAL TRIAL: NCT01481428
Title: Delivering HIV Risk Reduction Services in Treatment Court
Brief Title: Reducing High Risk Behavior in Treatment Court
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #1002; R01DA030257 (NIH)
Record Dates: First submitted 2011-11-18; First posted 2011-11-29 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance Abuse; HIV
Keywords: High risk behavior; Drug court clients; Substance abuse; HIV intervention; Treatment Court Clients
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention Control (Active Comparator)
  Interventions: Behavioral: Attention Control
- Computer-facilitated HIV intervention (Experimental)
  Interventions: Behavioral: Computer-facilitated HIV intervention

INTERVENTIONS:
Behavioral: Computer-facilitated HIV intervention — Individuals assigned to the experimental condition will complete the self-directed CARE HIV intervention during each of their first three sessions. The 20 minute intervention sessions involve several components including a brief risk assessment, review of identified risks, structured skill building videos, and the development of a risk prevention action plan. Because of the adaptive nature of the CARE program, the content of each session will be tailored to address the current risks of the participant. While the main focus of the intervention is on risk, individuals who report being HIV infected will receive a referral to treatment if they are not currently receiving medical care and their session will address, among other things, adherence to HIV care.
  Arms: Computer-facilitated HIV intervention
Behavioral: Attention Control — Life skills training DVDs that match the duration of the anticipated experimental condition. The DVDs address topics such as positive listening skills, anger management, and stress reduction.
  Arms: Attention Control

SUMMARY:
This study will be the first to examine the efficacy of using a brief, computerized HIV risk reduction intervention in treatment courts.

DETAILED DESCRIPTION:
Four hundred consenting treatment drug court participants will be randomly assigned to either an HIV intervention group (n = 200) or an attention control group. All clients will attend their regularly scheduled status hearings which are scheduled approximately every six weeks. Clients in the HIV intervention group will receive a brief computerized, self-administered HIV risk reduction intervention following each of their first three status hearings. Clients in the attention control condition will view a series of educational life-skill videos of matched length following each of their first three status hearings. The primary outcome will be engagement in high risk behaviors as measured by the Risk Assessment Battery (RAB). Secondary HIV-related outcomes will include: (1) rate of HIV testing, (2) condom procurement, and (3) self-reported condom use. Tertiary outcomes related to treatment court compliance will include: (1) drug court graduation, (2) urinalysis-confirmed drug abstinence, (3) case management attendance, and (4) satisfaction with case management. In addition, we will conduct preliminary cost and cost-effectiveness analyses on the delivery of the brief computerized HIV intervention. Assessments will be conducted at baseline and 9- and 15-months post admission.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years of age;
2. be charged with a non-violent felony offense
3. have no more than two prior non-violent convictions or diversionary opportunities
4. be willing to participate in the treatment court program for at least 12 months
5. be in need of treatment for substance abuse or dependence as assessed by case management.

Exclusion Criteria:

* Elderly subjects and those with medical problems will be included in the research as long as they do not have any physical or psychiatric condition that would impede their ability to give competent consent to research participation or to understand the research instruments.
* Those individuals who are intoxicated, cognitively impaired, or psychiatrically unstable when approached will not be included; however, such individuals may subsequently be included if the disqualifying condition subsides.
* Spanish speaking only individuals.
* Client remanded to jail or residential treatment facilities at the time of Treatment Court enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Engagement in high risk behaviors | 15 month follow-up
  Measured by the Risk Assessment Battery (RAB)

SECONDARY OUTCOMES:
Rate of HIV testing | 15 month follow-up
Condom Procurement | 15 month follow-up
Self-reported Condom Use | 15 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David S Festinger, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- Philadelphia Treatment Court, Philadelphia, Pennsylvania, United States